CLINICAL TRIAL: NCT04266340
Title: Effects of Different Premedication on Preoperative Sedation and Postoperative Agitation in Children Undergoing Ophthalmic and Otorhinolaryngologic Operations
Brief Title: Different Premedication in Pediatric Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20180341
Record Dates: First submitted 2020-01-13; First posted 2020-02-12 (Actual); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Agitation
MeSH Terms: conditions — Psychomotor Agitation | interventions — Dexmedetomidine; Midazolam; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo (Placebo Comparator): no premedication
  Interventions: Drug: Saline
- oralmidazolam (Experimental): 0.5 mg/kg oral midazolam group
  Interventions: Drug: midazolam
- intravenous midazolam (Experimental): 0.05 mg/kg intravenous injection midazolam group
  Interventions: Drug: midazolam
- dexmedetomidine (Experimental): 2.5µg/kg intranasal dexmedetomidine group
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: dexmedetomidine — 2.5µg/kg intranasal dexmedetomidine group
  Arms: dexmedetomidine
Drug: midazolam — 0.5mg/kg oral midazolam
  Arms: oralmidazolam
Drug: midazolam — 0.05mg/kg intravenous injection midazolam
  Arms: intravenous midazolam
Drug: Saline — no premedication
  Arms: placebo

SUMMARY:
The investigators studied the effects of intranasal dexmedetomidine compared with oral midazolam with different doses for premedication in children. One hundred and twenty children aged between 2 and 12 years were randomly allocated to one of four groups:2.5µg/kg intranasal dexmedetomidine group ; 0.5mg/kg oral midazolam group;0.05 mg/kg intravenous injection midazolam group; no premedication group.

Sedation levels 10, 20, and 30min after premedication were evaluated using a 5-point sedation scale. A 4-point emotional state score was used to evaluate participators when they were separated from their parents and their response to intravenous cannulation or facemask application. Agitation scores (Pediatric Anesthe-sia Emergence Delirium [PAED] scale) and POV were assessed in the postanesthetic care unit (PACU).Times to endotracheal tube or laryngeal mask airway removal, discharge from the PACU and patients' satisfaction degree were also assessed.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* a recent history of upper respiratory tract infection, a known allergy to dexmedetomidine or midazolam, inability to understand the consent process or parental refusal.

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 320 (Actual)
Dates: Start 2020-12-13 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Sedation | 10 minutes after premedication
  1. Rarely awake, needs shaking or shouting to wake up
  2. Asleep, eyes closed, wakes up when called softly or lightly touched
  3. Sleepy but eyes open spontaneously
  4. Awake
  5. Agitated
Sedation | 20 minutes after premedication
  1. Rarely awake, needs shaking or shouting to wake up
  2. Asleep, eyes closed, wakes up when called softly or lightly touched
  3. Sleepy but eyes open spontaneously
  4. Awake
  5. Agitated
Sedation | 30 minutes after premedication
  1. Rarely awake, needs shaking or shouting to wake up
  2. Asleep, eyes closed, wakes up when called softly or lightly touched
  3. Sleepy but eyes open spontaneously
  4. Awake
  5. Agitated
Emotional state | 0 minutes after they were separated from their parents
  1. Calm
  2. Apprehensive, not smiling, tentative behaviour, withdrawn
  3. Crying
  4. Thrashing, crying with movement of arms and legs, resisting
Emotional state | 0 minutes after intravenous cannulation
  1. Calm
  2. Apprehensive, not smiling, tentative behaviour, withdrawn
  3. Crying
  4. Thrashing, crying with movement of arms and legs, resisting
Emotional state | 0 minutes after facemask application
  1. Calm
  2. Apprehensive, not smiling, tentative behaviour, withdrawn
  3. Crying
  4. Thrashing, crying with movement of arms and legs, resisting

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology, The Eye, Ear, Nose and Throat Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiao H, Chen J, Lv P, Ye Z, Lu Y, Li W, Jia J. Efficacy of premedication with intravenous midazolam on preoperative anxiety and mask compliance in pediatric patients: a randomized controlled trial. Transl Pediatr. 2022 Nov;11(11):1751-1758. doi: 10.21037/tp-22-161. PMID 36506775